CLINICAL TRIAL: NCT07015190
Title: A Randomized, Phase 3, Open-label Study of Neoadjuvant Darovasertib in Subjects With Primary Non-metastatic Uveal Melanoma (OptimUM-10)
Brief Title: Neoadjuvant Darovasertib in Primary Uveal Melanoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IDEAYA Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDE196-010
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Uveal Melanoma
Keywords: Uveal Melanoma; Plaque Brachytherapy; Enucleation; Neoadjuvant; Darovasertib; IDE 196; Ocular Melanoma; Choroidal Melanoma; Ophthalmology; Ocular Oncology; Melanoma; Protein Kinase C; GNAQ; GNA11
MeSH Terms: conditions — Uveal Melanoma; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Darovasetib followed by definitive primary local therapy (i.e., PB, proton beam radiation, or enucleation)
  Interventions: Drug: Darovasertib
- Control Arm (Active Comparator): Immediate Primary Local therapy
  Interventions: Procedure: Primary Local Therapy

INTERVENTIONS:
Drug: Darovasertib — Dosed orally, twice daily (28-day/ cycle
  Other Names: IDE 196
  Arms: Treatment Arm
Procedure: Primary Local Therapy — Plaque Brachytherapy or Enucleation
  Arms: Control Arm

SUMMARY:
This is a Phase 3, randomized, multi-center, open-label study of neoadjuvant darovasertib in subjects with primary non-metastatic uveal melanoma (OptimUM-10)

DETAILED DESCRIPTION:
The study is divided into 2 cohorts of patients with primary uveal melanoma requiring either plaque brachytherapy or enucleation.

In cohort 1, patients in the treatment arm will receive neoadjuvant darovasertib followed by plaque brachytherapy compared to immediate plaque brachytherapy (control arm).

In cohort 2, the treatment arm will receive neoadjuvant darovasertib followed by definitive primary local therapy (i.e., plaque brachytherapy, proton beam radiation, or enucleation). Subjects in the control arm will go onto immediate enucleation.

Subjects will then receive primary local therapy following neoadjuvant darovasertib.

All patients will be followed for up to 3 years to assess longer term outcomes such as vision and tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Primary non-metastatic uveal melanoma
* Able and willing to provide written, informed consent before initiation of any study-related procedures, and in the opinion of the Investigator, to comply with all study requirements
* ECOG 0 or 1
* Adequate organ function

Exclusion Criteria:

* Previous treatment for UM
* Evidence of metastatic UM
* Attributes that necessitate enucleation regardless of response to therapy
* Evidence of progressive secondary underlying ocular disease that would confound longitudinal VA assessments
* Presence of a malignant disease other than the one being treated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: To demonstrate that the proportion of subjects with vision loss is lower for subjects in the Treatment Arm vs the Control Arm | Approximately 3 years
  Loss of Best Corrected Visual Acuity (BCVA) of ≥ 15 letters using Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA
Cohort 2: To demonstrate the ability to salvage the eye and prevent enucleation in the Treatment Arm | Approximately 2 years
  Eye preservation rate

CONTACTS AND LOCATIONS:
Locations (75):
- United States (27):
  - Mayo Clinic Scottsdale - PPDS, Scottsdale, Arizona
  - UCSD Moores Cancer Center, La Jolla, California
  - University of California Irvine Medical Center, Orange, California
  - Stanford Comprehensive Cancer Center, Palo Alto, California
  - Kaiser Permanente-Riverside Medical Center, Riverside, California
  - University of Colorado Hospital, Aurora, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Wilmer Eye Institute, Baltimore, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - W Kellogg Eye Center, Ann Arbor, Michigan
  - The Cancer and Hematology Centers of West Michigan (CHCWM), Grand Rapids, Michigan
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - TIERING Percentiles, Omaha, Nebraska
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center - 1275 York Ave, New York, New York
  - Cole Eye Institute-9500 Euclid Ave, Cleveland, Ohio
  - Ohio State Eye and Ear Institute, Columbus, Ohio
  - Jefferson Health Honickman Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Southeastern Retina Associates-Hixson, Hixson, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Austin Retina Associates - Central, Austin, Texas
  - Texas Retina Associates - Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center-5323 Harry Hines Blvd, Dallas, Texas
  - Augusta Health, Center for Cancer and Blood Disorders, Fishersville, Virginia
  - University of Wisconsin Health, Madison, Wisconsin
- Australia (2):
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - The Alfred Hospital, Melbourne, Victoria
- Austria (3):
  - LKH-Universitätsklinikum Graz, Graz
  - Universitätsklinikum Innsbruck, Innsbruck
  - Universitätsklinikum AKH Wien, Vienna
- Belgium (2):
  - Cliniques Universitaires Saint-Luc - PPDS, Brussels
  - UZ Leuven - PPDS, Leuven
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Ustredni vojenska nemocnice - Vojenska fakultni nemocnice Praha, Prague, Prague, Czechia
- Denmark (2):
  - Rigshospitalet, Copenhagen O, Capital
  - Aarhus Universitetshospital, Aarhus, Central Jutland
- East Tallinn Central Hospital-Pärnu road 104, Tallinn, Harju, Estonia
- France (4):
  - CHU de Nice-Hôpital Pasteur, Nice, Alpes-Maritimes
  - Centre Retine Gallien - Bordeaux, Bordeaux, Gironde
  - CHU de Rennes - Hôpital Pontchaillou, Rennes, Ille-et-Vilaine
  - Institut Curie - Hôpital de Paris, Paris, Paris
- Germany (9):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Städtisches Klinikum Dessau, Dessau, Saxony-Anhalt
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - Universitätsklinikum Giessen und Marburg - Marburg (UKGM), Marburg
  - Universitätsklinikum Würzburg, Würzburg
- PAGNI-University General Hospital of Heraklion, Heraklion, Irakleio, Greece
- Israel (2):
  - The Chaim Sheba Medical Center - PPDS, Ramat Gan, Central District
  - Hadassah Medical Center - PPDS, Jerusalem, Jerusalem
- Italy (6):
  - Istituto Nazionale Tumori IRCCS Fondazione Giovanni Pascale, Napoli, Campania
  - ASST Fatebenefratelli Sacco - Ospedale Luigi Sacco, Milan, Milan
  - Azienda Ospedaliera di Perugia - Ospedale Santa Maria della Misericordia, Perugia, Perugia
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliera di Perugia - Ospedale Santa Maria della Misericordia, Pisa
  - Fondazione Policlinico Universitario A Gemelli - Rome - PPDS, Rome
- Erasmus MC, Rotterdam, South Holland, Netherlands
- Poland (3):
  - Uniwersytecki Szpital Kliniczny w Poznaniu- Dluga 1/2, Poznan, Greater Poland Voivodeship
  - WIM-PIB, Centralny Szpital Kliniczny MON, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne w Gdansku - Debinki 7, Gdansk, Pomeranian Voivodeship
- Spain (6):
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid, Valladolid
  - Hospital Universitario Virgen Macarena, Seville
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Universitätsspital Zürich, Zurich
- United Kingdom (2):
  - Clatterbridge Cancer Centre - Liverpool - NWCRN - PPDS, Metropolitan Borough of Wirral, Merseyside
  - University College Hospital, London

IPD SHARING:
Plan to Share IPD: No